CLINICAL TRIAL: NCT05309096
Title: Evaluation of the Validity and Reliability of the Walking Adaptability Ladder Test (WAL-K) for Children in Children With Cerebral Palsy
Brief Title: Validity and Reliability of the WAL-K Test
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Taşvuran Horata, PhD; Assistant Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 2022/141
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Palsy; Gait Disorders in Children
Keywords: cerebral palsy; gait
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adapting the environment in which a child with Cerebral Palsy lives or adapting himself according to the environment facilitates independence in daily life activities. There is a need for practical performance tests to evaluate the gait adaptation of children with cerebral palsy in the clinic. However, no study has been found to evaluate gait adaptation in children with cerebral palsy. Therefore, the aim of the study is to evaluate the validity and reliability of the WALK test, which was previously developed for children with special learning disabilities, in individuals with cerebral palsy.

DETAILED DESCRIPTION:
According to the International Classification of Functioning, Disability, and Health, physical, social, and behavioral environmental factors; can affect a child's disability, activity limitations, and participation. Adapting the environment in which a child with Cerebral Palsy lives or adapting himself according to the environment facilitates independence in daily life activities. There is a need for practical performance tests to evaluate the gait adaptation of children with cerebral palsy in the clinic. However, no study has been found to evaluate gait adaptation in children with cerebral palsy. Therefore, the aim of the study is to evaluate the validity and reliability of the WALK test, which was previously developed for children with special learning disabilities, in individuals with cerebral palsy. The study will be conducted by Afyonkarahisar University Faculty of Health Sciences.

ELIGIBILITY:
Inclusion Criteria:

* 6-18 years of age;
* Diagnosed with Diparetic, Hemiparetic or Quadriparetic cerebral palsy;
* GMFCS value being ≤3.
* Communication Function Classification System (CFCS) for individuals with Cerebral Palsy ≤3.
* Children with a Modified Ashworth Scale (MASH) ≤ 3 for lower extremity muscles
* Ability to follow verbal commands
* Ability to recognize colors or numbers
* Able to walk ≥10 meters independently with or without an assistive device (orthotics or walking aid)

Exclusion Criteria:

* Presence of serious hearing, vision or cognitive problems,
* Nerve block injection or orthopedic surgery in the last 6 months (such as Botox injection or muscle lengthening surgery)
* Joint contracture

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will consist of children diagnosed with diparetic, hemiparetic, quadriparetic cerebral palsy with a functional level of 1, 2, or 3 according to Gross Motor Function Classification System (GMFCS) in Afyonkarahisar Special Education and Rehabilitation Center in Afyonkarahisar province.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
WAL-K test | 15 minutes
  The WAL-K test evaluates gait adaptation ability in children. A 10 meter long ladder is used for the test. The test is performed in two different conditions: taking only one step or taking two steps towards a target. The individual is video-recorded for the scoring of the test. Scoring records the total time (in seconds) and the total number of errors (tapping a stick, taking the wrong number of steps on a target, or missing a target) to complete the ladder back and forth. A combination score of time and errors is determined (0.5 s penalty is added to the elapsed time for each error). For the test, 1 trial and two formal tests are applied. The highest of the combination scores of the 2 formal tests is determined as the test result.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL TAŞVURAN HORATA, PhD, Principal Investigator — AFSU
Locations (1):
- Emel Taşvuran Horata, Afyonkarahisar, Turkey (Türkiye)